CLINICAL TRIAL: NCT03388957
Title: Evaluating of Oral Propranolol Effect on Managing Anxiety of Dental Extractions in Children: A Randomized Controlled Clinical Trial
Brief Title: Oral Propranolol for Reducing Pediatric Dental Patients Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UDDS-Pedo-02-2017
Record Dates: First submitted 2017-12-18; First posted 2018-01-03 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Extrusion of Tooth
MeSH Terms: interventions — Propranolol; Midazolam

STUDY DESIGN:
Intervention Model Description: Three groups, with 20 children in each group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propranolol (Experimental): Patients in this group will be given Propranolol 0.5 mg/Kg orally.
  Interventions: Drug: Propranolol
- Midazolam (Experimental): Patients in this group will be given Midazolam 0.5 mg/Kg orally.
  Interventions: Drug: Midazolam
- Propranolol and Midazolam (Experimental): Patients in this group will be given Propranolol and Midazolam with a dose of 0.5 mg/Kg orally for each drug.
  Interventions: Drug: Propranolol; Drug: Midazolam

INTERVENTIONS:
Drug: Propranolol — This drug will be given before the extraction procedure
  Arms: Propranolol; Propranolol and Midazolam
Drug: Midazolam — This drug will be given before the extraction procedure
  Arms: Midazolam; Propranolol and Midazolam

SUMMARY:
Evaluating anxiety, heart rate and behavior during dental extractions after oral dose of either Propranolol, Midazolam or a combination of both in uncooperative pediatric patients.

DETAILED DESCRIPTION:
Use of 0.5 mg/kg of Propranolol or a combination of Propranolol and Midazolam for the first time to manage uncooperative pediatric dental patients anxiety, comparing with Midazolam by evaluating anxiety, heart rate and behavior during administration of local anesthesia and extraction.

ELIGIBILITY:
Inclusion Criteria:

* High to extreme fear of tooth or molar anesthesia and removal (Frankl: Definitely negative).
* Scoring more than 19 points on MCDAS(f).
* Healthy pediatric patients (ASA I) aging 8-10 years.
* Indication for primary tooth or molar extraction.
* Fasting if indicated (severe gag reflex).
* Airway assessment (Mallampati and tonsillar hypertrophy).

Exclusion Criteria:

* Asthma or any other obstructive pulmonary disease.
* Cardiac failure.
* Cardiac arrhythmia.
* Renal failure.
* Diabetes.
* Current use of another ß-adrenoreceptor antagonist.
* Current use of anxiolytic or antidepressant medication.
* Currently in psychotherapy for dental anxiety.
* Systolic blood pressure <100 mmHg.
* Diastolic blood pressure <60 mmHg.
* Active Upper respiratory infection.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety-1 levels | (1) five minutes before medication, (2) 30 minutes post-extraction
  Anxiety-1 levels will be evaluated using self-reported faces anxiety scale (also called 'modified child dental anxiety scale). Scale name: Modified Child Dental Anxiety Scale (MCDAS):
  1. Relaxed/Not worried. (Better outcome)
  2. Very slightly worried.
  3. Fairly worried.
  4. Worried a lot.
  5. Very worried. (Worse outcome)
Change in Anxiety-2 levels | (1) 45 minutes after medication, while applying local anesthesia, (2) after 10 minutes of applying the anesthesia and during tooth extraction.
  Anxiety-2 levels will be measured using Observational Venham Anxiety Scale
  Major Issues: 1) Will be measured in 2 phases:
  * 45 minutes after medication, while applying local anesthesia.
  * While extracting the tooth. "Venham Anxiety Scale": 0. Relaxed. (Better outcome)
    1. Uneasy.
    2. Tense.
    3. Reluctant.
    4. Interference.
    5. Out of contact. (Worse outcome)
Change in heart rate | (1) 5 minutes before medication, (2) 45 minutes after medication, while applying local anesthesia, (3) after 10 minutes of applying the anesthesia and during tooth extraction, (4) 30 minutes following extraction
  using Finger Pulse Oximeter

SECONDARY OUTCOMES:
Change in Behavior | (1) 45 minutes after medication, while applying local anesthesia, (2) after 10 minutes of applying the anesthesia and during tooth extraction
  using Observational Frankl Scale "Frankl Scale":
  1. Definitely negative. (Worse outcome)
  2. Negative.
  3. Positive.
  4. Definitely positive. (Better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Abu Bakr, DDS, Principal Investigator — MSc student in Pedodontics, University of Damascus Dental School, Damascus, Syria; Mohamed Altinawi, DDS MSc PhD, Study Chair — Professor of Pedodontics, University of Damascus Dental School, Damascus, SYRIA; Youssef Latifeh, MD MSc Phd, Study Director — Professor and Head of the Psychiatry Department, Damascus Univesrity, Damascus, Syria
Locations (1):
- Department of Peadodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cote CJ, Wilson S; AMERICAN ACADEMY OF PEDIATRICS; AMERICAN ACADEMY OF PEDIATRIC DENTISTRY. Guidelines for Monitoring and Management of Pediatric Patients Before, During, and After Sedation for Diagnostic and Therapeutic Procedures: Update 2016. Pediatrics. 2016 Jul;138(1):e20161212. doi: 10.1542/peds.2016-1212. PMID 27354454
- [Background] Gazal G, Fareed WM, Zafar MS, Al-Samadani KH. Pain and anxiety management for pediatric dental procedures using various combinations of sedative drugs: A review. Saudi Pharm J. 2016 Jul;24(4):379-85. doi: 10.1016/j.jsps.2014.04.004. Epub 2014 Apr 26. PMID 27330369
- [Background] Heaton LJ, McNeil DW, Milgrom P. Propranolol and D-cycloserine as adjunctive medications in reducing dental fear in sedation practice. SAAD Dig. 2010 Jan;26:27-35. PMID 20151608
- [Background] LeCompte MT, Rae L, Kahn SA. A survey of the use of propranolol in burn centers: Who, what, when, why. Burns. 2017 Feb;43(1):121-126. doi: 10.1016/j.burns.2016.07.007. Epub 2016 Aug 27. PMID 27575676
- [Background] Steenen SA, van Wijk AJ, van der Heijden GJ, van Westrhenen R, de Lange J, de Jongh A. Propranolol for the treatment of anxiety disorders: Systematic review and meta-analysis. J Psychopharmacol. 2016 Feb;30(2):128-39. doi: 10.1177/0269881115612236. Epub 2015 Oct 20. PMID 26487439